CLINICAL TRIAL: NCT04665960
Title: Expert Statements on Infection Control in Intensive Care Unit for Severe Acute Respiratory Syndrome Coronavirus 2
Brief Title: Infection Control for Severe Acute Respiratory Syndrome Coronavirus 2
Acronym: IC-COVID-19
Status: Completed | Type: Observational
Sponsor: NMC Specialty Hospital (Other)
Responsible Party: Principal Investigator, Prashant Nasa, Head Critical Care Medicine, NMC Specialty Hospital
Other Study IDs: NMCSpecialtyH
Record Dates: First submitted 2020-12-09; First posted 2020-12-14 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Covid19; SARS-CoV Infection; SARS Pneumonia; Coronavirus Infection; Infection
Keywords: Infection Control; Intensive care unit; SARS-CoV-2; COVID-19
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome; Coronavirus Infections; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators aim to develop expert consensus statements on infection control management of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in intensive care units (ICU).

DETAILED DESCRIPTION:
The COVID-19 pandemic has resulted in a considerable change in the infection control protocols in the hospitals, especially ICU. The ICU management of these patients requires robust infection control measures in order to prevent cross-transmission of SARS-CoV-2 (to healthcare workers (HCWs) and other patients) and hospital acquired bacterial or fungal infections. The understanding of epidemiological characteristics of SARS-CoV-2 and pathophysiology of coronavirus disease 2019 (COVID-19) along with evidence on transmission of SARS-COV-2 in controlled healthcare-setting is still evolving. The mode of transmission of SARS-CoV-2 is airborne, through droplets or fomites. Respiratory interventions performed in these patients in ICU, such as non-invasive ventilation, high flow nasal oxygen or tracheal intubation are considered to be aerosol generating procedures and may lead to airborne transmission of SARS-CoV-2. In the absence of the robust evidence, there are no specific recommendations available on infection control of SARS-CoV-2 in ICU.

The objective of this study is to achieve consensus statements on the infection control management of SARS-CoV-2 in ICU.

The whole process of this study will be done in the form of three-four rounds of Google Forms-based Delphi surveys. The survey questionnaire, will be prepared by the investigators after systematic search of available literature and concern areas in the infection control of SARS-CoV-2 in ICU. The objective is to achieve consensus statements on the infection control management of SARS-CoV-2 in ICU.

The survey questionnaire is divided into five sections: 1.Design and engineering 2.Health-care workers and visitors 3. Personal protective equipment 4. Patient and procedures 5. Disinfection and sterilisation.

The majority of these questionnaire statements are to be rated on Likert scale and others have multiple choices. The participating experts comments and feedback will be collected through comment section after each question in round one. All the subsequent surveys will be iterative and the experts can give their opinion in each round using either open text or directly to steering group of investigators.

ELIGIBILITY:
Inclusion criteria for participants Health care professionals involved in the management of COVID-19 patients with publications and expertise in infectious disease, infection control, sepsis, respiratory failure or public health.

Exclusion Criteria:

* Those who do not accept the invitation or not meeting any of the inclusion criteria.

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 40 global experts in infectious disease, infection control, sepsis, respiratory failure or public health and involved in the management of COVD-19 will be invited to participate in study through e-mail with final expected participation of 35-40 experts.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2021-04-25 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Consensus using participating experts opinions. | 30 days
  For statements with responses on an ordinal 7-point Likert scale, 'agreement' is defined as a score of 5-7, 'neutral' by a score of 4 and 'disagreement' by a score of 1-3. Consensus is defined as achieved when >70% of the experts voted for a given option in Likert scale statement. Median and interquartile range (IQR) were used to describe the central tendency and dispersion of responses. For multiple-choice questions (MCQs), consensus is defined as achieved if >80% of the experts voted for a particular option.
  Stability in the responses will be assessed from round two onwards. Stability will be assessed between the two concluding rounds for each statement, using the non-parametric chi square (χ2) test. p < 0·05 is considered as a significant variation or unstable.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Myatra, MD, Principal Investigator — Tata Memorial Hospital, Mumbai, India
Locations (1):
- NMC Specialty Hospital, Dubai, United Arab Emirates

REFERENCES:
- [Background] Odor PM, Neun M, Bampoe S, Clark S, Heaton D, Hoogenboom EM, Patel A, Brown M, Kamming D. Anaesthesia and COVID-19: infection control. Br J Anaesth. 2020 Jul;125(1):16-24. doi: 10.1016/j.bja.2020.03.025. Epub 2020 Apr 8. PMID 32307115
- [Background] Wax RS, Christian MD. Practical recommendations for critical care and anesthesiology teams caring for novel coronavirus (2019-nCoV) patients. Can J Anaesth. 2020 May;67(5):568-576. doi: 10.1007/s12630-020-01591-x. Epub 2020 Feb 12. PMID 32052373
- See also: World Health Organisation (WHO). Infection prevention and control guidance - (COVID-19). Updated September 11, 2020. — https://www.who.int/westernpacific/emergencies/covid-19/technical-guidance/infection-prevention-control